CLINICAL TRIAL: NCT00574015
Title: The Comparison of Supraperiosteal Nerve Block With Opiate Analgesia in Alleviating the Pain of Toothache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Wayne Triner, Professor Emergency Medicine, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2200; 2200
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2010-09

CONDITIONS: Toothache
Keywords: toothache; regional anesthesia; emergency department
MeSH Terms: conditions — Toothache; Emergencies | interventions — oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral (Active Comparator): administration of oral analgesia
  Interventions: Drug: hydrocodone/acetaminophen
- Dental Block (Experimental): Administration of supraperiosteal nerve block to effected tooth
  Interventions: Drug: bupivacaine (supraperiosteal nerve block)

INTERVENTIONS:
Drug: hydrocodone/acetaminophen — oral hydrocodone 10 mg/acetaminophen 650 mg
  Other Names: Lortab; Vicodin
  Arms: oral
Drug: bupivacaine (supraperiosteal nerve block) — Administration of Bupivacaine 0.5% 2 ml adjacent to tooth root
  Other Names: Marcaine
  Arms: Dental Block

SUMMARY:
This study will compare the degree of pain control provided by two techniques for persons with toothache in an emergency department. The two techniques include;

* standard oral narcotic pain medication
* numbing the tooth with local anesthetic by needle injection

DETAILED DESCRIPTION:
Background: Toothache is a common complaint among patients presenting to the emergency department. There are two commonly employed methods of alleviating this severe form of pain. Oral opioid analgesia is the most commonly utilized strategy for treating this pain. However, many emergency physicians and dentists employ a local anesthetic technique known as supraperiosteal nerve block. This study will compare the relative efficacy of these techniques.

Patients meeting enrollment criteria will be randomized to either receive a supraperiosteal nerve block or oral hydrocodone 10 mg/acetaminophen 650 mg. They will otherwise be managed identically. Reduction of pain scores between entry and 30 minutes post intervention will be compared as well as numeric pain scores obtained by phone contact 24 hours later. Secondary outcomes will include the proportion of individuals from each group filling prescriptions for pain medication and the number of pain pills taken.

ELIGIBILITY:
Inclusion Criteria:

* Involvement of a single tooth
* Percussive tenderness of the crown of the suspect tooth

Exclusion Criteria:

* Age younger than 18 years
* Women who are breast feeding
* Allergy or intolerance to hydrocodone, bupivacaine or acetaminophen
* Pregnancy
* Involvement of multiple teeth
* Pain resulting from pericoronitis.
* Pain resulting from dental trauma occurring less than 90 days prior
* Pain of more than 96 hours duration
* Facial or neck swelling or tenderness
* Alteration in phonation
* Cognitive impairment
* Concurrent use of opiate analgesics
* Impairment of liver function
* Consumption of more than 4 grams of acetaminophen in the past 24 hours.
* Patients who are visually impaired.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
VAS determination of pain at 30 minutes following intervention | 30 minutes

SECONDARY OUTCOMES:
Numeric scale report or pain Number of prescribed analgesic pills taken | 24-36 hours following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wayne R Triner, DO, MPH, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center Hospital, Albany, New York, United States